CLINICAL TRIAL: NCT04254575
Title: Smartphone-based Digital Phenotyping to Detect High-risk Affect States in Body Dysmorphic Disorder (BDD)
Brief Title: Understanding Daily Changes in BDD Risk Using Smartphones
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hilary Weingarden, Psychologist, Massachusetts General Hospital
Other Study IDs: 2019P002041
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Body Dysmorphic Disorders
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- body dysmorphic disorder (BDD): Adults with a current primary diagnosis of body dysmorphic disorder (BDD)
  Interventions: Other: None, observational study only (no interventions)

INTERVENTIONS:
Other: None, observational study only (no interventions) — None, observational study only (no interventions)

SUMMARY:
Body dysmorphic disorder (BDD) is associated with high risk for suicide attempts (22-28%) and substance use disorders (49%), underscoring the importance of accurate, real-time risk detection in BDD. This study aims to use smartphone-based digital phenotyping to develop and validate unobtrusive, time-sensitive, and ecologically valid measures of key risk factors for suicide and substance misuse in BDD: negative affect states. As next steps, this research can be extended to detect risk transdiagnostically, with the goal of enabling just-in-time interventions to target suicide and substance misuse across psychiatric illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >=18
* Current primary diagnosis of BDD
* BDD severity >= moderate
* Living in US
* English proficiency
* Owns an Android or iOS (Apple) smartphone
* Has regular Wifi-enabled internet access for data downloads

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a current primary diagnosis of body dysmorphic disorder (BDD) within the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Self-reported anxiety intensity, rated from 1 (very slightly or not at all) to 5 (extremely) | 3 months
  Ecological momentary assessment (EMA) of anxiety intensity, where higher scores indicated more severe anxiety.
Self-reported shame intensity, based on Positive and negative affect scale (PANAS) shame item, rated from 1 (very slightly or not at all) to 5 (extremely) | 3 months
  Ecological momentary assessment (EMA) of shame intensity, where higher scores indicate more severe shame.
Self-reported negative affect intensity, based on Positive and negative affect scale (PANAS) negative affect items (averaged), rated from 1 (very slightly or not at all) to 5 (extremely) | 3 months
  Ecological momentary assessment (EMA)-rated general negative affect intensity, where higher scores indicate more severe negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Weingarden, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Weingarden H, Jaroszewski AC, Armey M, Hoeppner BB, Armstrong CH, Onnela JP, Wilhelm S. Predicting concurrent and short-term desire and intent to attempt suicide among people with body dysmorphic disorder using ecological momentary assessment of anxiety and shame. J Psychopathol Clin Sci. 2025 Oct 6:10.1037/abn0001054. doi: 10.1037/abn0001054. Online ahead of print. PMID 41051851
- [Derived] Weingarden H, Meng X, Armey M, Onnela JP, Jaroszewski A, Armstrong CH, Wilhelm S. Predicting the strength of next-day negative emotion states in body dysmorphic disorder using passive smartphone data: An intensive longitudinal assessment study. Internet Interv. 2025 May 15;40:100833. doi: 10.1016/j.invent.2025.100833. eCollection 2025 Jun. PMID 40486130